CLINICAL TRIAL: NCT00884624
Title: Evaluation of the PillCam™ Colon Capsule -2 System
Status: Completed | Type: Observational
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: MA-200
Record Dates: First submitted 2009-04-20; First posted 2009-04-21 (Estimated); Last update posted 2019-07-31 (Actual); Status verified 2010-03

CONDITIONS: Bowel Diseases
Keywords: Bowel Diseases
MeSH Terms: conditions — Intestinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A: Subjects that are indicated for colonoscopy, who are suspected or known to suffer from large bowel diseases.

SUMMARY:
The purpose of this study is to evaluate the ability of the PillCam Colon Capsule 2 to detect polyps and other pathologies in the colon.

DETAILED DESCRIPTION:
Standard evaluation of subjects with suspected colon diseases includes endoscopic imaging by colonoscopy and radiology testing such as: air-contrast barium enema, abdominal/pelvic CT, or virtual colonoscopy.

The Given® Diagnostic System offers an alternative approach for endoscopic visualization of the colon. Advantages of the Given® Diagnostic System include the elimination of the need for conscious sedation, the minimally invasive, painless nature of the exam, and the ability to pursue normal daily activities immediately following the procedure . Furthermore, compared to standard colonoscopy, the Given® Diagnostic System may be more readily accepted by the subjects, thereby improving subjects' willingness to undergo a diagnostic evaluation of the colon and comply with colorectal cancer screening recommendations.

The PillCam™ SB capsule (formerly M2A® Capsule) that was cleared by the FDA- in August 2001 for small bowel evaluation has been ingested to date by more than 500,000 people worldwide and is well accepted by patients and physicians as well as the professional societies. However, adequate visualization of the colon cannot be achieved with the standard PillCam™ SB capsule because of the anatomical and physiological properties of the colon which are significantly different than the small bowel. Moreover, other issues that limit the evaluation of the colonic mucosa by the standard PillCam™ SB procedure include an unsatisfactory level of colon cleanliness and slow progression of the PillCam™ SB capsule through the colon during the desired examination time. Therefore, the development and introduction of a specially designed, customized colon capsule combined with a dedicated capsule colonoscopy procedure protocol will allow for more efficient evaluation of the colonic mucosa. This is expected to improve the capability of the Given® Diagnostic System to detect colonic pathologies and to serve as a diagnostic and screening tool for colonic disease. To date, several clinical studies have been conducted with PillCam™ Colon Endoscope 1(PCCE-1) system. The new development of PillCam Colon Endoscope 2 (PCCE-2) is primarily aimed to increase sensitivity and specificity for polyp detection.

Further details of the PillCam™ Colon Capsule Endoscope (PCCE-2) can be found in the device description section.

This study is designed to evaluate the performance of the new version of colon capsule and its performance in detecting lesions in the colon as compared to conventional colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Subject is between the ages of 18-57 years.
* Subject is able and agrees to sign the Informed Consent Form
* Subject was referred to colonoscopy for at least one of the following reasons:

  * Colorectal cancer screening
  * Clinical symptoms such as: rectal bleeding, hematochezia, melena, positive FOBT, recent change of bowel habits, or diarrhea/constipation of recent onset.
  * Positive findings in the colon on a GI radiographic study
  * Personal history of colorectal cancer (CRC) or adenomatous polyps and at least 5 years since last conventional colonoscopy
  * Positive findings in the colon
  * Personal history of polyps that were removed at least 5 years ago (5 years and more)

Exclusion Criteria:

* Subject has dysphagia
* Subject has congestive heart failure
* Subject has renal insufficiency
* Subject has Nephrotic syndrome
* Subject has Cirrhosis
* Subject is known or is suspected to suffer from intestinal obstruction.
* Subject is taking NSAID medication
* Subject suffers from hypertension and is taking one or more of the following medications used for control of hypertension: diuretics, ACE inhibitors, Angiotensin II blockers
* Chronic use of laxatives
* Subject has a cardiac pacemakers or other implanted electro medical devices.
* Women who are either pregnant or nursing at the time of screening, who intend to be during the study period, or are of child-bearing potential and do not practice medically acceptable methods of contraception.
* Subject is expected to undergo MRI examination within 7 days after ingestion of the capsule.
* Subject has had prior abdominal surgery of the gastrointestinal tract other than uncomplicated procedures that would be unlikely to lead to bowel obstruction based on the clinical judgment of the investigator.
* Subject has any condition, which precludes compliance with study and/or device instructions.
* Age < 18 years or under parent guardian
* Age>57 years
* Subject suffers from life threatening conditions
* Subject is currently participating in another clinical study
* Subject has known slow gastric emptying time
* Subject is allergic or contraindicated to any of the study medications

Ages: 18 Years to 57 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Subjects that are indicated for colonoscopy, who are suspected or known to suffer from large bowel diseases.
Sampling Method: Non-Probability Sample
Enrollment: 255 (Actual)
Dates: Start 2009-03; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Accuracy parameters of PCCE-2 in detecting colonic polyps as compared to conventional colonoscopy | Within 7 Days
Assessment of colon cleansing level at different colon segments | Within 7 days
Distribution of capsule excretion time | Within 7 Days
Percent of excreted capsules up to 10 hours post capsule ingestion. | Within 7 Days
Number, type and severity of adverse events | WithIn 7 days

SECONDARY OUTCOMES:
Accuracy parameters of PCCE-2 in detecting colonic lesions as compared to conventional colonoscopy | within 7 days
Capsule transit time within stomach, small bowel and colon | within 7 days
Number of polyps and sizes at different colon segments detected by capsule | within 7 days
Number of polyps and sizes at different colon segments detected by conventional colonoscopy | within 7 days
RAPID video reading time | Within 7 days
Conventional colonoscopy duration including: total time, insertion time, and withdrawal time see my comment above (at the objective section) | Within 7 Days
Assessment of the RAPID video | Within 7 Days
Patient questionnaire | Within 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Rami Eliakim, Prof., Principal Investigator — Rambam Health Care Campus
Locations (5):
- Israel (5):
  - Hillel Yaffe Hospital, Hadera
  - Rambam - Medical center, Haifa
  - Bikkur Holim Hospital, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center, Petah Tikva